CLINICAL TRIAL: NCT04125147
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Investigation of MONTAGE in Adults With Spinal Deformity Undergoing Pedicle Subtraction Osteotomy
Brief Title: Clinical Investigation of MONTAGE in Adults With Spinal Deformity Undergoing Pedicle Subtraction Osteotomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Abyrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20182341
Record Dates: First submitted 2019-10-09; First posted 2019-10-14 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Fused Vertebrae; Ankylosing Spondylitis; Sagittal Deformities; Thoracolumbar Kyphosis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Montage Bone Hemostat (Experimental): Use of Montage Settable Resorbable Hemostatic bone putty on the cut surfaces of bleeding bone at the osteotomy site
  Interventions: Device: Experimental: Montage Bone Hemostat
- Standard of Care: No bone hemostat (No Intervention): Use of no bone hemostat on the cut surfaces of bleeding bone at the osteotomy site

INTERVENTIONS:
Device: Experimental: Montage Bone Hemostat — Use of Montage bone hemostat on the cut surfaces of bone at the osteotomy site
  Arms: Montage Bone Hemostat

SUMMARY:
This study evaluates the difference in postoperative bleeding between two study groups, FDA cleared MONTAGE Settable Resorbable Hemostatic Bone Putty and standard of care (no bone hemostat) during pedicle subtraction osteotomy procedures.

DETAILED DESCRIPTION:
Pedicle Subtraction osteotomy (PSO) is a surgical option for treating several spinal deformities. It has been utilized in alignment disorders of the fused spine, in the lumbar spine to treat large sagittal deformities and in patients with ankylosing spondylitis with thoracolumbar kyphotic deformity.

PSO typically results in substantial loss of blood (as much as 2L) with a significant portion of the loss likely occurring at the osteotomy surfaces post-surgically. The control of peri-operative blood loss is considered a critical issue by spine surgeons. A variety of methods have been proposed for the reduction of blood loss during or immediately after spine surgery, including preoperative use of erythropoietin, autologous blood, cell salvage, intra-operative controlled hypotension, and the use of anti-fibrinolytic drugs. Bone hemostats have traditionally not been part of the standard of care to promote hemostasis probably because most traditional options (e.g., bone wax) are nonabsorbable and thus might interfere with fusion at the osteotomy site.

MONTAGE is a settable (hardening) bioabsorbable polymer and hydroxyapatite/beta tricalcium phosphate based putty, used in the control of bleeding from bone during spine, orthopedic, craniomaxillofacial, thoracic and other surgical procedures, and has been FDA cleared.

ELIGIBILITY:
Inclusion Criteria:

* Presence of spinal deformity requiring a PSO at a single site level, such as for patients with thoracolumbar kyphotic deformity, sagittal imbalance, and spinal global malalignment.
* Non-smokers (have proven to quit smoking for at least 6 months prior to surgery) and current smokers.
* Female subjects of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence). A pregnancy test at the Week 0 visit must be administered, and must be negative, for inclusion into the study.
* Subject understands and is willing to participate in the clinical study and can comply with required visits and the follow-up regimen.
* Subject has read and signed the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

* Subjects whose spinal deformity is deemed by the investigator to be of such severity that a possible surgical intervention would be either harmful or not warranted.
* Subjects with morbid obesity (i.e. a Body Mass Index [BMI] ≥ 40).
* Subjects who have a known allergy to the components of MONTAGE.
* Subjects who are non-mobile (i.e. not ambulatory, or have significant impairment of their mobility making them completely bedridden).
* Subjects who, in the opinion of the investigator, show evidence of infection, cellulitis, and/or osteomyelitis.
* Subjects with abnormally low platelets, abnormal coagulation parameters, or with documented bleeding disorders, including a prior history of excessive bleeding during surgery.
* Subjects with a history of a malignancy, not in remission for five years or more, or a newly diagnosed malignancy, treated with cytotoxic therapies or radiation therapy.
* Subjects on any investigational drug(s) within 30 days preceding randomization (i.e. Week 0); or subject or physician anticipates use of any of these therapies by the subject during the course of the study.
* Subjects with:

  (i) Alcohol abuse as recorded by an average daily intake of > 4 units in females, > 5 units in males (i.e. 1 oz. of spirit, glass of wine, or can of beer per unit).

(ii) Drug abuse as evidenced by the subject's use of illegal drugs or prescription drugs that have not been prescribed for him/her.

* Subjects with one or more medical conditions, as determined by medical history, including renal, hepatic, hematologic, active auto-immune or immune diseases that, in the opinion of the Investigator, would make the subject an inappropriate candidate for this study.
* Subjects with a history of osteoporosis, as defined by imaging, or on medication for osteoporosis or documented fracture of fragility (Hip fracture, osteoporotic compression fracture, distal radius fracture). If there are any concerns these may be arbitrated by the study PI.
* Subject has previously participated in any MONTAGE trial.
* Subjects who are unable to understand the aims and objectives of the trial and/or unwilling to return for the follow-up examinations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Hemostasis | Week 0
  The primary objective of this study is to evaluate the difference in postoperative bleeding between two study groups, FDA cleared MONTAGE and standard of care (no bone hemostat), and the extent to which any transfusion is needed.
Hemostasis | Week 0
  The primary objective of this study is to evaluate the difference in postoperative bleeding between two study groups, FDA cleared MONTAGE and standard of care (no bone hemostat), with blood loss is measured through drop in hematocrit (HCT).
Hemostasis | Week 0
  The primary objective of this study is to evaluate the difference in postoperative bleeding between two study groups, FDA cleared MONTAGE and standard of care (no bone hemostat) as wound drain output, if utilized.

SECONDARY OUTCOMES:
PSO Stability | 1-year and 2-years post surgery
  The secondary objective is the stability of the construct, as measured by whether the correction has maintained stability at 1-year and 2-years post surgery. Each incidence of instability will be categorized as belonging to one of the following groups: 1) hardware malplacement, 2) loosening or dislodgement, 3) nonunion or nonfusion with hardware fracture 4) nonunion or nonfusion without hardware fracture and 5) perihardware fracture.

CONTACTS AND LOCATIONS:
Overall Officials: William Lavelle, MD, Principal Investigator — SUNY Upstate
Locations (1):
- Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cogniet A, Aunoble S, Rigal J, Demezon H, Sadikki R, Le Huec JC. Clinical and radiological outcomes of lumbar posterior subtraction osteotomies are correlated to pelvic incidence and FBI index : Prospective series of 63 cases. Eur Spine J. 2016 Aug;25(8):2657-67. doi: 10.1007/s00586-016-4424-5. Epub 2016 Feb 10. PMID 26861730
- [Background] Liu H, Yang C, Zheng Z, Ding W, Wang J, Wang H, Li S. Comparison of Smith-Petersen osteotomy and pedicle subtraction osteotomy for the correction of thoracolumbar kyphotic deformity in ankylosing spondylitis: a systematic review and meta-analysis. Spine (Phila Pa 1976). 2015 Apr 15;40(8):570-9. doi: 10.1097/BRS.0000000000000815. PMID 25868095
- [Background] Bridwell KH. Decision making regarding Smith-Petersen vs. pedicle subtraction osteotomy vs. vertebral column resection for spinal deformity. Spine (Phila Pa 1976). 2006 Sep 1;31(19 Suppl):S171-8. doi: 10.1097/01.brs.0000231963.72810.38. PMID 16946635
- [Background] Bridwell KH, Lewis SJ, Lenke LG, Baldus C, Blanke K. Pedicle subtraction osteotomy for the treatment of fixed sagittal imbalance. J Bone Joint Surg Am. 2003 Mar;85(3):454-63. doi: 10.2106/00004623-200303000-00009. PMID 12637431
- [Background] Hyun SJ, Kim YJ, Rhim SC. Spinal pedicle subtraction osteotomy for fixed sagittal imbalance patients. World J Clin Cases. 2013 Nov 16;1(8):242-8. doi: 10.12998/wjcc.v1.i8.242. PMID 24340276
- [Background] Lee EI, Chao AH, Skoracki RJ, Yu P, DeMonte F, Hanasono MM. Outcomes of calvarial reconstruction in cancer patients. Plast Reconstr Surg. 2014 Mar;133(3):675-682. doi: 10.1097/01.prs.0000438061.46290.33. PMID 24263391
- [Background] Cheng L, Ye F, Yang R, Lu X, Shi Y, Li L, Fan H, Bu H. Osteoinduction of hydroxyapatite/beta-tricalcium phosphate bioceramics in mice with a fractured fibula. Acta Biomater. 2010 Apr;6(4):1569-74. doi: 10.1016/j.actbio.2009.10.050. Epub 2009 Nov 5. PMID 19896564
- [Background] Pripatnanont P, Praserttham P, Suttapreyasri S, Leepong N, Monmaturapoj N. Bone Regeneration Potential of Biphasic Nanocalcium Phosphate with High Hydroxyapatite/Tricalcium Phosphate Ratios in Rabbit Calvarial Defects. Int J Oral Maxillofac Implants. 2016 Mar-Apr;31(2):294-303. doi: 10.11607/jomi.4531. PMID 27004276
- [Background] Koshiyama H, Yamazaki K. Absorbable sternal pins improve sternal closure stability within a small deviation. Gen Thorac Cardiovasc Surg. 2015 Jun;63(6):331-4. doi: 10.1007/s11748-015-0533-z. Epub 2015 Feb 27. PMID 25720972
- [Background] Baumgart D, Herbon G, Borowski A, de Vivie ER. Primary closure of median sternotomy with interposition of hydroxyapatite blocks. A new approach in pediatric cardiac surgery. Eur J Cardiothorac Surg. 1991;5(7):383-5. doi: 10.1016/1010-7940(91)90057-q. PMID 1832549
- [Background] Barbanti Brodano G, Griffoni C, Zanotti B, Gasbarrini A, Bandiera S, Ghermandi R, Boriani S. A post-market surveillance analysis of the safety of hydroxyapatite-derived products as bone graft extenders or substitutes for spine fusion. Eur Rev Med Pharmacol Sci. 2015 Oct;19(19):3548-55. PMID 26502842
- [Background] Yi S, Rim DC, Park SW, Murovic JA, Lim J, Park J. Biomechanical Comparisons of Pull Out Strengths After Pedicle Screw Augmentation with Hydroxyapatite, Calcium Phosphate, or Polymethylmethacrylate in the Cadaveric Spine. World Neurosurg. 2015 Jun;83(6):976-81. doi: 10.1016/j.wneu.2015.01.056. Epub 2015 Mar 10. PMID 25769482

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT04125147/Prot_SAP_001.pdf